CLINICAL TRIAL: NCT00486109
Title: A Study Assessing an Injection Port for Administration of Insulin
Brief Title: A Prospective, Randomized, Parallel Crossover Study Demonstrating Subject Wearability and Usability of the I-Port Injection Port
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patton Medical Devices (Industry)
Collaborators: Medstar Health Research Institute (Other); Valeritas, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PTN 012.1
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: I-Port(TM) Injection Port

SUMMARY:
This study investigated wearability and usability of the I-PORT™ Injection Port (I-PORT™), a new disposable injection port through which prescribed medication is injected subcutaneously from a standard syringe or pen. Additional investigation compared subject opinion towards using the I-PORT™ device compared to standard injection therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 14-70 years of age, with type 1 and type 2 diabetes mellitus for a minimum of six (6) months
* Subjects must be utilizing a regimen of at least two (2)injections daily of either Novolin®, Humulin®, NovoLog®, Humalog® or Apidra® and no more than one (1) injection of Lantus® daily using a standard syringe or insulin pen
* Current regimen of intensified insulin therapy (defined as separate injections of basal and prandial insulin with at least three (3) insulin injections per day) for a minimum of three (3) months
* Body Mass Index <35 kg/m2
* HbA1c ≤ 10 %
* If medications (other than oral anti-diabetic agents) in addition to insulin are taken at screening, the subject must be on a stable regimen as defined by continued use of the same dose of each medication for a period of at least three (3) months prior to study enrollment
* Subjects must be willing to provide written informed consent

Exclusion Criteria:

* Use of Continuous Subcutaneous Insulin Infusion (CSII) at any time within the preceding three (3) months
* History or current diagnosis of chronic diseases which in the view of the PI would interfere with adequate involvement in and completion of the requirements of the study
* Use of short term or chronic steroids within two (2) months of entry into the study or likelihood that same might be required during the conduct of the study
* Use of hydrochlorthiazide at doses >25 mg daily
* Use of beta-blocker drugs
* Regular pre-prandial doses of SC insulin >30 IU per meal
* Intake of any drug or herbal preparation which, in the evaluation of the PI, may interfere with the interpretation of clinical study results or that is known to cause clinically relevant interference with insulin action, glucose utilization or ability to detect or recover from hypoglycemia (e.g., systemic steroids)
* History of known hypersensitivity to plastics or polymers
* Treatment with any investigational drug within two (2) months prior to enrollment or during this study
* Progressive fatal disease
* History of malignancy within five (5) years of study entry(other than basal cell carcinoma)
* Evidence of severe secondary complications of diabetes(neuropathy, nephropathy as evidenced by creatinine >1.5 mg/dL for females or >1.8 mg/dL for males, grade III or IV retinopathy or severe peripheral vascular disease)
* Evidence of gastroparesis, orthostatic hypotension or hypoglycemia unawareness (autonomic neuropathy)
* Myocardial infarction or stroke within the preceding six (6)months
* Positive hepatitis B (HBsAg) and/or hepatitis C (Hep C AB)serology and/or positive HIV serology
* History or presence of clinically significant cardiovascular, hepatic (as evidenced by ALT or AST >3 times the upper limit of normal), gastrointestinal, neurological or infectious disorders capable of altering the absorption, metabolism or elimination of drugs, or constituting a significant risk factor when using the study device
* Anemia (hemoglobin levels <11 g/dL for females or <12 g/dL for males)
* Pregnancy, lactation, or intention to become pregnant
* Female subjects of childbearing potential practicing inadequate birth control (adequate birth control is defined as using oral
* Regular alcohol intake greater than 18 units*/week, or subjects unwilling to stop alcohol for the duration of the study (* 1 unit = 8 g ethanol, ¼ liter of beer or 1 glass wine or 1 ounce of spirits)
* PI or clinical site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted
* A lack of compliance (including the inability to maintain a minimum of 75% compliance with study device administration) or other reasons, which in the opinion of the PI may preclude the participation of the subject in the study

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-10; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Glycosylated albumin levels | 7 weeks

SECONDARY OUTCOMES:
Participants' satisfaction evaluated with standard quality of life questionnaires and adverse events related to the study device including incidents of erythema > 2cm diameter, incidence of induration > 1cm dimater and incidence of suppuration. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sherwyn Schwartz, M.D., Principal Investigator — Diabetes and Glandular Disease Clinic; Bruce Bode, M.D., Principal Investigator — Atlanta Diabetes Associates; Thomas Blevins, M.D., Principal Investigator — Texas Diabetes & Endocrinology; Stephen Aronoff, M.D., Principal Investigator — Research Institute of Dallas; Claire Baker, M.D., Principal Investigator — Diabetes and Endocrine Associates
Locations (5):
- United States (5):
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Diabetes and Endocrine Associates, Omaha, Nebraska
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas